CLINICAL TRIAL: NCT02867813
Title: A Multicenter, Open-label, Single-arm, Extension Study to Assess Long-term Safety of Evolocumab Therapy in Patients With Clinically Evident Cardiovascular Disease
Brief Title: Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With Elevated Risk Open-label Extension
Acronym: FOURIER OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130295; 2015-004780-36 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-08-16 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Dyslipidemia
Keywords: High Cholesterol; Treatment for high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- evolocumab (AMG 145) (Experimental): All subjects are randomized to a single arm and will receive evolocumab 140mg every two weeks (Q2W) or 420mg monthly (QM) according to subject's preference.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — subjects will receive evolocumab 140 mg every 2 weeks (Q2W) or 420 mg monthly (QM), according to the subject's preference.

SUMMARY:
The primary clinical hypothesis is that long-term exposure of evolocumab will be safe and well tolerated in subjects with clinically evident atherosclerotic cardiovascular disease (CVD).

DETAILED DESCRIPTION:
This is a multicenter, open-label extension study designed to assess the long-term safety of evolocumab in subjects who completed the FOURIER study,which is a randomized placebo-controlled study of evolocumab in subjects with clinically evident atherosclerotic CVD on stable effective statin therapy. Eligible subjects at sites participating in FOURIER OLE who have signed the FOURIER OLE informed consent may be enrolled at the completion of FOURIER study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent before initiation of any study-specific activities/procedures
* Subject has completed FOURIER (Study 20110118) while still receiving assigned investigational product.

Exclusion Criteria:

* Investigational product was permanently discontinued during FOURIER for any reason, including an adverse event or serious adverse event
* Subject is currently receiving treatment in another investigational device or drug study, or ended treatment on another investigational device or drug study(ies) within less than 4 weeks. Other investigational procedures while participating in this study are excluded
* Subject is not likely to be available to complete protocol-required study visits or procedures and/or to comply with required study procedures to the best of the subject's and investigator's knowledge
* Subject has a history or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Subject has a known sensitivity to any of the active substances or excipients (eg, sodium acetate) to be administered during dosing
* Female subject is pregnant or breastfeeding or is planning to become pregnant or planning to breastfeed during treatment with evolocumab and within 15 weeks after the end of treatment with evolocumab
* Female subjects of childbearing potential who are not willing to use an acceptable method(s) of effective birth control during treatment with evolocumab and for an additional 15 weeks after the end of treatment with evolocumab are excluded

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5035 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (184):
- United States (139):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Banning, California
  - Research Site, Long Beach, California
  - Research Site, Oceanside, California
  - Research Site, Oxnard, California
  - Research Site, Palm Springs, California
  - Research Site, Roseville, California
  - Research Site, San Diego, California
  - Research Site, San Pedro, California
  - Research Site, Tarzana, California
  - Research Site, Torrance, California
  - Research Site, Valley Village, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Ponte Vedra Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Addison, Illinois
  - Research Site, Belleville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Jerseyville, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Hammond, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Natchitoches, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Newton, Massachusetts
  - Research Site, Grandville, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, West Seneca, New York
  - Research Site, Williamsville, New York
  - Research Site, Calabash, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Willoughby, Ohio
  - Research Site, Pryor, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Moncks Corner, South Carolina
  - Research Site, North Myrtle Beach, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Layton, Utah
  - Research Site, West Jordan, Utah
  - Research Site, Burke, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Federal Way, Washington
  - Research Site, Seattle, Washington
  - Research Site, Green Bay, Wisconsin
- Czechia (10):
  - Research Site, Brno
  - Research Site, Jihlava
  - Research Site, Liberec
  - Research Site, Mohelnice
  - Research Site, Ostrava
  - Research Site, Ostrava-Dubina
  - Research Site, Prague
  - Research Site, Pribram VIII
  - Research Site, Přerov
  - Research Site, Znojmo
- Hungary (3):
  - Research Site, Békéscsaba
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
- Poland (26):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nysa
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Pszczyna
  - Research Site, Puławy
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Staszów
  - Research Site, Świdnik
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zamość
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- Slovakia (2):
  - Research Site, Košice
  - Research Site, Svidník
- Research Site, Zaporizhzhya, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] O'Donoghue ML, Giugliano RP, Wiviott SD, Atar D, Keech A, Kuder JF, Im K, Murphy SA, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Sabatine MS. Long-Term Evolocumab in Patients With Established Atherosclerotic Cardiovascular Disease. Circulation. 2022 Oct 11;146(15):1109-1119. doi: 10.1161/CIRCULATIONAHA.122.061620. Epub 2022 Aug 29. PMID 36031810
- [Background] Gaba P, O'Donoghue ML, Park JG, Wiviott SD, Atar D, Kuder JF, Im K, Murphy SA, De Ferrari GM, Gaciong ZA, Toth K, Gouni-Berthold I, Lopez-Miranda J, Schiele F, Mach F, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Giugliano RP, Sabatine MS. Association Between Achieved Low-Density Lipoprotein Cholesterol Levels and Long-Term Cardiovascular and Safety Outcomes: An Analysis of FOURIER-OLE. Circulation. 2023 Apr 18;147(16):1192-1203. doi: 10.1161/CIRCULATIONAHA.122.063399. Epub 2023 Feb 13. PMID 36779348
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension of study 20110118 (NCT01764633). Eligible participants were enrolled after the completion of the 20110118 study. 5035 participants were enrolled at 195 centers in Czech Republic, Hungary, Poland, Russia, Slovakia, Ukraine, and the United States from 02 September 2016 to 17 March 2022.
Pre-assignment Details: 5035 participants were enrolled and 5031 of those participants received study drug.
Groups:
- Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study: Participants in the parent study who received placebo subcutaneous injections either Q2W or QM, and received evolocumab 140 mg every 2 weeks Q2W or 420 mg monthly QM in the open label extension, according to the participant's preference.
- Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study: Participants in the parent study who received evolocumab subcutaneous injections either Q2W or QM, and received evolocumab 140 mg Q2W or 420 mg QM in the open label extension according to the participant's preference.
Period: Overall Study
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study
Started | 2535 | 2500
Completed | 2084 | 2090
Not Completed | 451 | 410
Not completed — Withdrawal by Subject | 57 | 56
Not completed — Decision by Sponsor | 7 | 7
Not completed — Lost to Follow-up | 91 | 78
Not completed — Missing | 2 | 1
Not completed — Death | 294 | 268

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants is made up of all of the participants that received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Total
Number analyzed (Participants) | 2532 | 2499 | 5031
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (8.4) | 62.4 (8.5) | 62.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 638 | 622 | 1260
  Male | 1894 | 1877 | 3771
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 63 | 118
  Not Hispanic or Latino | 2477 | 2436 | 4913
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 5 | 2 | 7
    Asian | 9 | 21 | 30
    Black or African American | 111 | 117 | 228
    Native Hawaiian or Other Pacific Islander | 5 | 4 | 9
    White | 2392 | 2345 | 4737
    Multiple | 4 | 4 | 8
    Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: All adverse event summaries for the primary analysis of the primary endpoint (OLE study period only) included all treatment-emergent events reported on the Event electronic case report form (eCRF), including CEC positively reviewed events and disease-related events.
Time Frame: Up to 5 years
Population: OLE Safety Analysis Set which included all participants who received at least 1 dose of open-label evolocumab in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study
Number analyzed (Participants) | 2532 | 2499
Participants | 2144 | 2084

2. Secondary Outcome: Percent Change of Low-density Lipoprotein Cholesterol (LDL-C) From Baseline at Each Scheduled Visit
Time Frame: Week 12, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, Week 192, Week 216, Week 260
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study
Number analyzed (Participants) | 2532 | 2499
Percent Change
  Week 12: number analyzed (Participants) | 2438 | 2408
  Week 12 | -55.93 (33.73) | -58.43 (30.64)
  Week 24: number analyzed (Participants) | 2444 | 2410
  Week 24 | -56.69 (33.58) | -58.38 (31.52)
  Week 48: number analyzed (Participants) | 2378 | 2370
  Week 48 | -58.52 (33.66) | -59.05 (33.06)
  Week 72: number analyzed (Participants) | 2327 | 2325
  Week 72 | -56.35 (33.73) | -56.90 (33.14)
  Week 96: number analyzed (Participants) | 2281 | 2275
  Week 96 | -55.70 (33.72) | -56.62 (33.36)
  Week 120: number analyzed (Participants) | 2228 | 2233
  Week 120 | -53.37 (36.77) | -54.89 (35.99)
  Week 144: number analyzed (Participants) | 2156 | 2185
  Week 144 | -56.96 (32.82) | -57.38 (32.34)
  Week 168: number analyzed (Participants) | 2113 | 2151
  Week 168 | -56.49 (37.04) | -58.22 (34.60)
  Week 192: number analyzed (Participants) | 1583 | 1608
  Week 192 | -57.42 (35.43) | -58.81 (33.27)
  Week 216: number analyzed (Participants) | 1764 | 1753
  Week 216 | -54.68 (35.53) | -57.11 (32.89)
  Week 260: number analyzed (Participants) | 1882 | 1884
  Week 260 | -53.69 (37.51) | -56.63 (36.14)

3. Secondary Outcome: Percentage of Participants Who Achieved an LDL-C Level < 40 mg/dL
Time Frame: Week 12, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, Week 192, Week 216, Week 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once a Month (QM) in Parent Study
Number analyzed (Participants) | 2532 | 2499
Percentage of Participants
  Week 12: number analyzed (Participants) | 2438 | 2408
  Week 12 | 58.7 [56.7 to 60.6] | 61.4 [59.4 to 63.3]
  Week 24: number analyzed (Participants) | 2444 | 2410
  Week 24 | 60.2 [58.2 to 62.1] | 61.6 [59.7 to 63.5]
  Week 48: number analyzed (Participants) | 2378 | 2370
  Week 48 | 61.7 [59.8 to 63.7] | 61.9 [60.0 to 63.9]
  Week 72: number analyzed (Participants) | 2327 | 2325
  Week 72 | 59.7 [57.7 to 61.7] | 58.5 [56.5 to 60.5]
  Week 96: number analyzed (Participants) | 2281 | 2275
  Week 96 | 57.3 [55.3 to 59.3] | 59.9 [57.8 to 61.9]
  Week 120: number analyzed (Participants) | 2228 | 2233
  Week 120 | 54.6 [52.5 to 56.6] | 56.4 [54.4 to 58.5]
  Week 144: number analyzed (Participants) | 2156 | 2185
  Week 144 | 59.6 [57.6 to 61.7] | 60.4 [58.3 to 62.4]
  Week 168: number analyzed (Participants) | 2113 | 2151
  Week 168 | 60.9 [58.8 to 63.0] | 61.5 [59.4 to 63.5]
  Week 192: number analyzed (Participants) | 1583 | 1608
  Week 192 | 61.8 [59.4 to 64.1] | 62.3 [59.9 to 64.7]
  Week 216: number analyzed (Participants) | 1764 | 1753
  Week 216 | 56.0 [53.6 to 58.3] | 59.2 [56.9 to 61.5]
  Week 260: number analyzed (Participants) | 1882 | 1884
  Week 260 | 56.9 [54.6 to 59.1] | 59.2 [56.9 to 61.4]

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 5 years during the OLE study.
Description: All-Cause Mortality is reported for all enrolled participants. Serious and Other Adverse Events are reported for the Safety Analysis Set defined as all participants who received at least 1 dose of open-label evolocumab in the OLE study.
Groups:
- Placebo in Parent Study: Participants with Placebo in Parent Study
- Evolocumab in Parent Study: Participants with Evolocumab in Parent Study
Arm/Group | Placebo in Parent Study | Evolocumab in Parent Study
All-Cause Mortality (participants affected / at risk) | 309/2535 | 287/2500
Serious Adverse Events (participants affected / at risk) | 1077/2532 | 1045/2499
Other Adverse Events (participants affected / at risk) | 956/2532 | 959/2499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Parent Study (N=2532) | Evolocumab in Parent Study (N=2499)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 13 | 18
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 5 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Acute cardiac event (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 10 | 6
Acute left ventricular failure (Cardiac disorders) | 5 | 3
Acute myocardial infarction (Cardiac disorders) | 74 | 52
Angina pectoris (Cardiac disorders) | 56 | 52
Angina unstable (Cardiac disorders) | 49 | 37
Aortic valve disease (Cardiac disorders) | 1 | 1
Aortic valve disease mixed (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmic storm (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 57 | 47
Atrial flutter (Cardiac disorders) | 11 | 13
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 9 | 9
Atrioventricular block second degree (Cardiac disorders) | 4 | 5
Bradycardia (Cardiac disorders) | 8 | 9
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 16 | 13
Cardiac asthma (Cardiac disorders) | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 46 | 44
Cardiac failure acute (Cardiac disorders) | 21 | 17
Cardiac failure chronic (Cardiac disorders) | 13 | 23
Cardiac failure congestive (Cardiac disorders) | 37 | 40
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 5 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 2
Cardiovascular disorder (Cardiac disorders) | 4 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 3
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 41 | 30
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 4 | 5
Coronary artery stenosis (Cardiac disorders) | 8 | 4
Heart valve incompetence (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 5
Left ventricular failure (Cardiac disorders) | 8 | 4
Mitral valve incompetence (Cardiac disorders) | 1 | 3
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 25 | 20
Myocardial ischaemia (Cardiac disorders) | 15 | 11
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 2 | 2
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 7 | 8
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 8
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 4 | 6
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 4 | 3
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 17 | 14
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 2
Talipes (Congenital, familial and genetic disorders) | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
External ear disorder (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 2 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 4
Vertigo labyrinthine (Ear and labyrinth disorders) | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 3 | 0
Vestibular ataxia (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 11 | 8
Choroidal detachment (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Epiretinal membrane (Eye disorders) | 0 | 1
Eyelid bleeding (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Macular rupture (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 2
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 3 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 2 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal symptom (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal stenosis (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 5
Colitis ischaemic (Gastrointestinal disorders) | 2 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Colon dysplasia (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 4 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 1
Femoral hernia strangulated (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 2
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 2 | 0
Gastric volvulus (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 16
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 8 | 11
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 3 | 6
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 5 | 1
Pancreatitis acute (Gastrointestinal disorders) | 5 | 10
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 3
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 4
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 1
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 4
Subileus (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 6 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 8
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 5 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 15 | 7
Complication associated with device (General disorders) | 0 | 1
Death (General disorders) | 9 | 10
Exercise tolerance decreased (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 0 | 1
Implant site pain (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 6
Non-cardiac chest pain (General disorders) | 26 | 37
Pneumatosis (General disorders) | 1 | 0
Prosthetic cardiac valve stenosis (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Stent-graft endoleak (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 7 | 3
Sudden death (General disorders) | 10 | 6
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent occlusion (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 2
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 4
Cholecystitis acute (Hepatobiliary disorders) | 7 | 10
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 13 | 11
Chronic hepatic failure (Hepatobiliary disorders) | 2 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 1
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 2
Liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess bacterial (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acute endocarditis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 7 | 1
Appendicitis perforated (Infections and infestations) | 4 | 0
Arthritis bacterial (Infections and infestations) | 1 | 2
Arthritis infective (Infections and infestations) | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 8 | 10
COVID-19 (Infections and infestations) | 15 | 15
COVID-19 pneumonia (Infections and infestations) | 32 | 23
Cellulitis (Infections and infestations) | 17 | 20
Cholecystitis infective (Infections and infestations) | 1 | 1
Cholera (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Coccidioidomycosis (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 3 | 3
Cystitis klebsiella (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Diabetic foot infection (Infections and infestations) | 1 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 11 | 7
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 2
Eczema infected (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 2
Extradural abscess (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 3 | 5
Gastroenteritis (Infections and infestations) | 4 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1
Groin abscess (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 11 | 6
Intervertebral discitis (Infections and infestations) | 1 | 0
Joint abscess (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 2 | 0
Meningoencephalitis viral (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 6 | 2
Osteomyelitis acute (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Perihepatic abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 50 | 74
Pneumonia aspiration (Infections and infestations) | 4 | 5
Pneumonia bacterial (Infections and infestations) | 9 | 3
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 2 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 5 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rocky mountain spotted fever (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 14 | 23
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 3 | 3
Serratia infection (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 14 | 13
Urinary tract infection bacterial (Infections and infestations) | 3 | 3
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 7 | 4
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 2
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 2
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 10
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 6 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 2
Frostbite (Injury, poisoning and procedural complications) | 1 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 5 | 9
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 5
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 2
Pelvic organ injury (Injury, poisoning and procedural complications) | 0 | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 4
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 3 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 5
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 3
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 1
Squamous cell carcinoma antigen (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Troponin I increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 8 | 12
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Mineral deficiency (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee impingement syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 37 | 36
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 8
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 5
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 10
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Anal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign male reproductive tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign spleen tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer stage I, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage I, without cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phosphaturic mesenchymal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 16
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Vulval cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Basilar artery stenosis (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 2
Carotid artery disease (Nervous system disorders) | 2 | 3
Carotid artery occlusion (Nervous system disorders) | 1 | 2
Carotid artery stenosis (Nervous system disorders) | 11 | 10
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral ataxia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 5 | 2
Cerebral infarction (Nervous system disorders) | 4 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 25 | 20
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 2 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 8 | 2
Dizziness postural (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 4 | 1
Encephalopathy (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 2
Facial paralysis (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 3 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 2 | 3
Hemianopia (Nervous system disorders) | 0 | 1
Hemiparaesthesia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 18 | 27
Lacunar infarction (Nervous system disorders) | 1 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 3 | 1
Migraine (Nervous system disorders) | 2 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Moyamoya disease (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paresis cranial nerve (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral nerve lesion (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Phantom limb syndrome (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Post stroke epilepsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 2
Psychogenic seizure (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 4 | 0
Seizure (Nervous system disorders) | 1 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 19 | 14
Thalamic infarction (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 11 | 14
Vascular dementia (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 2 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 2
Vertebrobasilar stroke (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 2 | 0
Device failure (Product Issues) | 1 | 0
Device loosening (Product Issues) | 2 | 0
Device malfunction (Product Issues) | 0 | 2
Device mechanical issue (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Device power source issue (Product Issues) | 1 | 1
Device stimulation issue (Product Issues) | 0 | 1
Lead dislodgement (Product Issues) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 4
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 2 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 2
Major depression (Psychiatric disorders) | 1 | 1
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 9 | 3
Paranoia (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 25 | 30
Bladder stenosis (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 3 | 6
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 4
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 4 | 9
Nephropathy toxic (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal embolism (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 2
Renal haematoma (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 5
Urethral perforation (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 | 7
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1
Pelvic organ prolapse (Reproductive system and breast disorders) | 0 | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0
Uterine inflammation (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 23
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 25 | 30
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epiglottic mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Tissue expansion procedure (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 2
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 13 | 10
Aortic aneurysm rupture (Vascular disorders) | 3 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 7 | 10
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial perforation (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 3 | 7
Arteriovenous fistula (Vascular disorders) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1
Blue toe syndrome (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 4
Diabetic macroangiopathy (Vascular disorders) | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 5
Embolism arterial (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Giant cell arteritis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 20 | 10
Hypertensive crisis (Vascular disorders) | 3 | 4
Hypertensive emergency (Vascular disorders) | 1 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 7 | 5
Hypovolaemic shock (Vascular disorders) | 1 | 3
Iliac artery embolism (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 2
Intermittent claudication (Vascular disorders) | 1 | 2
Internal haemorrhage (Vascular disorders) | 1 | 1
Leriche syndrome (Vascular disorders) | 3 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 5 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 24 | 26
Peripheral artery aneurysm (Vascular disorders) | 4 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 3
Peripheral artery stenosis (Vascular disorders) | 1 | 3
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Peripheral circulatory failure (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 6 | 10
Peripheral vascular disorder (Vascular disorders) | 4 | 10
Peripheral venous disease (Vascular disorders) | 1 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 2 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 2
Subclavian artery embolism (Vascular disorders) | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Subclavian vein occlusion (Vascular disorders) | 1 | 0
Superior vena cava stenosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 4
Varicose vein (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous haemorrhage (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Parent Study (N=2532) | Evolocumab in Parent Study (N=2499)
Bronchitis (Infections and infestations) | 162 | 173
Nasopharyngitis (Infections and infestations) | 157 | 156
Upper respiratory tract infection (Infections and infestations) | 208 | 162
Diabetes mellitus (Metabolism and nutrition disorders) | 139 | 135
Arthralgia (Musculoskeletal and connective tissue disorders) | 144 | 138
Back pain (Musculoskeletal and connective tissue disorders) | 133 | 137
Hypertension (Vascular disorders) | 327 | 355

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT02867813/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02867813/SAP_001.pdf